CLINICAL TRIAL: NCT03084354
Title: Women's Experiences of Maternity Bladder Care
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 19544
Record Dates: First submitted 2017-03-07; First posted 2017-03-20 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Bladder Care
Keywords: pelvic floor; women's experiences; bladder care; pregnancy; labour; postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured interviews — Semi-structure interviews to gain a deep understanding of women's experiences of maternity bladder care. Interviews will last between thirty minutes to a couple of hours and they will be digitally recorded and transcribed verbatim.

SUMMARY:
Background.

Although a healthy urinary system is a vital aspect in every woman's life, bladder management is an aspect of maternity care, which is, or perceived as, being poorly managed by health care professionals. Furthermore, although the relationship between childbirth and bladder dysfunction is an incontestable fact very well documented in the medical literature, women's experiences of bladder care have not been recognized by the evidence, and therefore, no research has been developed to address this topic. This fact implies a limited level of awareness and degree of implication from women in this matter.

Research question.

What are women's experiences, perceptions and knowledge of bladder care during the antepartum, intrapartum and postpartum period?

Aim.

To explore women's experiences of bladder care during the antepartum, intrapartum and postpartum period.

Design.

Exploratory, descriptive research study.

Population.

Women who have given birth to a singleton, live, term baby between two weeks and six months prior the study, and who meet the inclusion and exclusion criteria.

Methods.

In-depth semi-structured interviews.

Sample.

A purposive sample of eight to sixteen women, with a heterogeneous representation of the different modes of birth, will be sought.

Recruitment.

Postnatal midwives will act as gatekeepers identifying potential participants and providing information packs. Other recruitment resources will include posters and a study website, which will be advertised at local maternity groups.

Data collection.

Semi-structure interviews to gain a deep understanding of women's experiences of maternity bladder care. Interviews will last between thirty minutes to a couple of hours and they will be digitally recorded and transcribed verbatim.

Data Analysis.

Framework analysis assisted by memoing technique.

Ethical considerations.

Ethical approval from the Sponsor and the Health Research Authority will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Women who have received antepartum, intrapartum and postpartum care at the designated hospital.
* Women who have given birth to a live singleton, term (37 to 42 weeks gestation) infant between two weeks and six months ago at the designated hospital.
* Women who have been identified and received the information pack by the named postnatal midwife. Alternatively, potential participants can also get included in the study after being self-referred through local maternity groups (posters, leaflets, (PDF file) webpages and study website).

Exclusion Criteria:

* Women and newborns with serious medical/life threatening conditions (pre-existing mental health, neurological, uro-genital conditions, pregnancy related complications and/or newborn related conditions, such us, preterm delivery, fetal abnormalities, admission to the neonatal unit and poor condition at birth).
* Women who have experienced a stillbirth, neonatal death or traumatic birth.
* Women who are not fluent in English, although Spanish participants will be included as the main researcher is fluent in both languages.
* Women under the age of eighteen.
* Women who are unable to be interviewed due to cognitive impairment or disabilities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The target population is women who have received antepartum, intrapartum and postpartum care at the designated hospital and have birthed a live singleton, term baby (37-42 weeks gestation) between two weeks to six months prior to the interview.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Women's experiences of bladder care during the antepartum, intrapartum and postpartum period | day 1
  Qualitative semi-structured interviews performed at one occasion where the participant describes her experience of bladder care during pregnancy, labour and after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ellen Kitson-Reynolds, Study Chair — University of Southampton; Veronica Blanco-Gutierrez, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: study website — https://bladdercarematernitystudy.wordpress.com